CLINICAL TRIAL: NCT01959646
Title: The Effect of Aged Garlic Extract Supplementation on the Immune System
Brief Title: The Effect of AGE on the Immune System
Acronym: EAGESIS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB201300529
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Immune Function; Aged Garlic Extract; Supplementation; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Group
  Interventions: Other: Standard for Groups; Dietary Supplement: Placebo
- Aged Garlic Extract Supplementation (Experimental): Aged Garlic Extract Supplementation Group
  Interventions: Dietary Supplement: Aged Garlic Extract Supplementation Group; Other: Standard for Groups

INTERVENTIONS:
Dietary Supplement: Aged Garlic Extract Supplementation Group — Subjects will be asked to consume three (3) capsules of 600 mg aged garlic extract (AGE) with food twice a day, for a total of 3.6 grams per day.
  Other Names: AGE
  Arms: Aged Garlic Extract Supplementation
Other: Standard for Groups — To assess for eligible study participants, the research team will use the Cholestech LDX® System (Alere™ Inc, Waltham, MA) to analyze finger-prick blood samples. This is an efficient and economical point of care testing for c-Reactive Protein (CRP), cholesterol and related lipids, and blood glucose, as diagnostic tools which provide information for immediate risk assessment and therapeutic monitoring of heart disease, inflammatory disorders and diabetes. Each finger prick will be treated individually.
Dietary Supplement: Placebo — Participants will be asked to consume three (3) placebo capsules with food twice a day.
  Arms: Placebo

SUMMARY:
This is a nutritional intervention study using healthy overweight/obese humans to investigate if a supplement made from aged garlic extract has an impact on immunity. Following a baseline blood draw, participants will consume the capsules (garlic or placebo) for 42 days, at which time a second blood draw will occur. Tests for immune function and inflammation will be performed on both the baseline and 42 day samples. The investigators anticipate that the immune functions and biomarkers that are inflammatory in an overweight/obese population will be returning to normal after 42 days of consumption of this supplement. The investigators predict that AGE supplementation will benefit immunity and improve function while reducing inflammation in a stressed population (inflamed obese).

DETAILED DESCRIPTION:
Healthy, overweight adults age 25 to 65 will be recruited, consented and screened for eligibility. To assess for eligible study participants, the investigators will use the Cholestech LDX® System (Alere™ Inc, Waltham, MA) to analyze finger-prick blood samples. This is an efficient and economical point of care testing for c-Reactive Protein (CRP), cholesterol and related lipids, and blood glucose, as diagnostic tools which provide information for immediate risk assessment and therapeutic monitoring of heart disease, inflammatory disorders and diabetes. Each finger prick will be treated individually. To this end, universal precautions such as hand washing, glove change, new lancet, etc. will be utilized for every finger prick throughout the assessment.

Eligible participants will be enrolled, and subsequently return, to provide a baseline blood draw, and given their random group assignment. Participants will be asked to consume three (3) capsules of 600 mg AGE or placebo with food twice a day, for a total of 3.6 grams per day. This dose was determined from previous studies that analyzed for cardiovascular risk factors. The supplementation (AGE and placebo) intervention will occur over 42 days, sometime between September 2013 and February 2013. Blood will be taken again at 42 days, two (2) hours after subjects have taken their capsules. A light breakfast will be offered after both fasting blood draws.

Peripheral blood mononuclear cells will be isolated from the blood at both blood draws and either used fresh, or cultured in autologous serum for 24 hours. Freshly isolated cells will be used to determine compliance (glutathione); population numbers of γδ T cells and monocytes and their function (activation); and mRNA expression of IL-6 and TNF-α. After 24 hours of stimulation with a broad based mitogen, culture medium will be harvested and assayed for IL-6, and TNF-α proteins. The cultured cells will be assayed for γδ T cell and monocyte function and for mRNA analysis of IL-6 and TNF-α gene expression. The serum obtained at both blood draws will be used in cultures as autologous serum and for assay of inflammatory biomarkers (C-reactive protein, IL-6, TNF-α, adiponectin and leptin). Compliance will also be determined by capsule count.

ELIGIBILITY:
Inclusion Criteria:

* ages 25-65
* BMI > or = to 30 kg/m2
* willing to discontinue dietary supplements
* cRP between 2 and 10 mg/L

Exclusion Criteria:

* medication for hypertension, high cholesterol, heart failure, angina, etc
* diagnoses of diabetes, metabolic syndrome, arthritis, severe allergies, or any other compromised immune condition
* blood pressure > 135/85 mmHg
* serum triglycerides > 150 mg/dl
* HDL cholesterol < 40 mg/dl for men or < 50 mg/dl for women
* fasting glucose > 110 mg/dl

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Markers of immune health | 6 weeks
  Number and function of gamma delta T-cells and monocytes

SECONDARY OUTCOMES:
Markers of inflammation | 6 weeks
  IL-6 and TNF alpha

OTHER OUTCOMES:
Serum antioxidant status (compliance) | 6 weeks
  Serum glutathione

CONTACTS AND LOCATIONS:
Overall Officials: Susan Percival, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Food Science & Human Nutrition Building, University of Florida, Gainesville, Florida
  - University of Florida, Gainesville, Florida

REFERENCES:
- [Derived] Xu C, Mathews AE, Rodrigues C, Eudy BJ, Rowe CA, O'Donoughue A, Percival SS. Aged garlic extract supplementation modifies inflammation and immunity of adults with obesity: A randomized, double-blind, placebo-controlled clinical trial. Clin Nutr ESPEN. 2018 Apr;24:148-155. doi: 10.1016/j.clnesp.2017.11.010. Epub 2018 Jan 3. PMID 29576354